CLINICAL TRIAL: NCT02144077
Title: A Randomized, Observer Blind, Multinational Phase III Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) in Comparison to Metvix® in the Treatment of Non-aggressive Basal Cell Carcinoma (BCC) With Photodynamic Therapy (PDT)
Brief Title: Safety and Efficacy Study for the Treatment of Non-Aggressive Basal Cell Carcinoma With Photodynamic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Collaborators: Accovion GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALA-BCC-CT008; 2013-003241-42 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-05-21 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Basal Cell Carcinoma (BCC)
Keywords: Photodynamic Therapy; PDT; non-aggressive BCC
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — BF-200 ALA; Aminolevulinic Acid; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF-200 ALA (Active Comparator): Topical application of BF-200 ALA gel containing 78 mg/g 5-aminolevulinic acid. Application of a 1 mm thick layer covering each lesion and 0.5 to 1 cm of surrounding margin.
  Interventions: Drug: BF-200 ALA
- methyl-aminolevulinate (Active Comparator): Topical application of Metvix creme containing 160 mg/g methyl-aminolevulinate. Application of a 1 mm thick layer covering each lesion and 0.5 to 1 cm of surrounding margin.
  Interventions: Drug: methyl-aminolevulinate

INTERVENTIONS:
Drug: BF-200 ALA — Topical treatment for photodynamic therapy combining drug application and subsequent illumination with a narrow spectrum light source (after 3 h of drug incubation)
  Other Names: Ameluz
  Arms: BF-200 ALA
Drug: methyl-aminolevulinate — Topical treatment for photodynamic therapy combining drug application and subsequent illumination with a narrow spectrum light source (after 3 h of drug incubation)
  Other Names: Metvix / Metvixia
  Arms: methyl-aminolevulinate

SUMMARY:
The aim of this study is to test the effectiveness and safety of the medicine Ameluz® (5-aminolevulinic acid) in comparison to methyl-aminolevulinate (MAL), used with photodynamic therapy (PDT), to treat thin, non-aggressive BCC (basal cell carcinoma).

DETAILED DESCRIPTION:
The treatment comprises of up to 2 PDT cycles, each with two PDT sessions one week apart.

If 12 weeks after the the second PDT all lesions are completely cleared the patient will enter the follow-up phase. In case of remaining lesions the patient will receive a second PDT cycle starting on the same day.

ELIGIBILITY:
Main Inclusion Criteria:

* Willing and able to sign informed consent form; obtained in writing before starting any study procedures
* Presence of 1-3 thin (≤2 mm thickness), clinically non-aggressive, primary BCC lesions (primary superficial, nodular, or mixed superficial/nodular) in the face/forehead, bald scalp, extremities and/or neck/trunk. Confirmation of non-aggressiveness and thickness of BCC through biopsies taken at screening for at least one lesion. Lesions non-eligible according to biopsy should timely be removed by surgery or cryotherapy
* Diameters of lesions should range between ≥0.5cm and ≤2cm; total maximal treated area is 10cm² (including 0.5-1.0cm margin surrounding each lesion)
* Target BCC lesions must be discrete and quantifiable and have to be located within 1-2 treatment areas
* Free of significant physical abnormalities (eg tattoos, dermatoses) in potential treatment area that may cause difficulty with examination or final evaluation
* Accept to abstain from extensive sunbathing and use of solarium during observer blind part. Patients with sunburn within treatment areas cannot be included until fully recovered
* Healthy patients and patients with clinically stable medical conditions, including, but not limited to controlled hypertension, diabetes mellitus type II, hypercholesterolemia, and osteoarthritis, will be permitted to be included in study if their medication is not prohibited by protocol
* Women of childbearing potential are permitted to participate in study only if they have a negative serum pregnancy test at screening and willingness to use a highly effective method of contraception during observer blind part

Main Exclusion Criteria:

* History of hypersensitivity to 5-ALA or any ingredient of BF-200 ALA, MAL or any ingredient of Metvix®, including arachis oil, or to peanut or soya
* Hypersensitivity to porphyrins
* Current treatment with immunosuppression therapy
* Presence of porphyria
* Presence of BCC lesions on embryonic fusion planes (H-zone)
* Presence of more than 3 BCCs
* Presence of malignant or benign tumors of the skin other than non-aggressive BCC within the treatment area (eg malignant melanoma, squamous cell carcinoma (SCC), aggressive BCC clinically diagnosed at screening) within the last 12 weeks
* Gorlin Syndrome or Xeroderma pigmentosum
* Presence of photodermatoses
* Treatment of lesions (actinic keratosis (AK), BCC, SCC, Bowens disease, melanoma) ≤12 weeks prior to first PDT, except physical treatments (eg cryosurgery, excision surgery) that will not be allowed ≤6 weeks prior to first PDT (Visit 2). Lesion(s) that seemed eligible clinically which could not be confirmed by biopsy, and which are located ≥10cm to an eligible lesion should timely be removed physically only
* Presence of inherited or acquired coagulation defect
* Start of intake of medication with hypericin or systemically-acting drugs with phototoxic or photoallergic potential within 8 weeks prior to screening
* Clinically relevant cardiovascular, hepatic, renal, neurologic, endocrine, or other major systemic disease making implementation of protocol or interpretation of study results difficult
* Evidence of clinically significant (CS), unstable medical conditions, eg:

  * Metastatic tumor or tumor with high probability of metastasis
  * Cardiovascular disease (New York Heart Association [NYHA] class III, IV)
  * Immunosuppressive condition
  * Hematologic, hepatic, renal, neurologic, or endocrine condition
  * Collagen-vascular condition
  * Gastrointestinal condition
* Topical treatment with 5-ALA or MAL outside treatment area during the observer blind part
* Any topical treatment including diclofenac and immunomodulatory agents (eg imiquimod, ingenol mebutate) 12 weeks prior to first PDT session and during observer blind part
* Any physical treatment during the observer blind part within treated target areas with exception of lesion(s) determined non-eligible by biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf M. Szeimies, Prof. Dr., Principal Investigator — Klinik fuer Dermatologie und Allergologie (Klinikum Vest - Knappschaftskrankenhaus), Recklinghausen, Germany; Colin Morton, Dr., Principal Investigator — Dermatology Department, Stirling Community Hospital, NHS Forth Valley, United Kingdom
Locations (1):
- Klinikum Vest GmbH, Recklinghausen, Westfalen-Lippe, Germany

REFERENCES:
- [Result] Morton CA, Dominicus R, Radny P, Dirschka T, Hauschild A, Reinhold U, Aschoff R, Ulrich M, Keohane S, Ekanayake-Bohlig S, Ibbotson S, Ostendorf R, Berking C, Grone D, Schulze HJ, Ockenfels HM, Jasnoch V, Kurzen H, Sebastian M, Stege H, Staubach P, Gupta G, Hubinger F, Ziabreva I, Schmitz B, Gertzmann A, Lubbert H, Szeimies RM. A randomized, multinational, noninferiority, phase III trial to evaluate the safety and efficacy of BF-200 aminolaevulinic acid gel vs. methyl aminolaevulinate cream in the treatment of nonaggressive basal cell carcinoma with photodynamic therapy. Br J Dermatol. 2018 Aug;179(2):309-319. doi: 10.1111/bjd.16441. Epub 2018 May 16. PMID 29432644
- See also: US National Library of Medicine National Institutes of Health — http://www.ncbi.nlm.nih.gov/pubmed/29432644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted in Germany and United Kingdom with a total of 24 sites who recruited patients.
  Enrollment of patients started (first patient enrolled) 28-Jan-2014.
Pre-assignment Details: Of the 394 patients screened in this study, 281 patients were randomized (138 patients to BF-200 ALA and 143 patients to methyl-aminolevulinate) and treated. 113 patients were excluded before randomization due to screening failure (104 patients), patient's decision (7 patients), and lost to FU and "other reason" (each 1 patient).
Groups:
- BF-200 ALA: Topical application of BF-200 ALA gel (78 mg/g 5-aminolevulinic acid). The dose of BF-200 ALA was up to 1 g per PDT session (depending on size and number of target lesions located on neck, trunk, extremities, face or scalp, no more than 2 illumination areas with a maximum area incl. margin of 10cm², and a film thickness of about 1mm). Up to 4 administrations of study treatment (i.e. PDT sessions: drug application and subsequent illumination with BF-RhodoLED after 3h of drug incubation) were applied. For all patients, PDT-1 was to be administered directly after randomization and PDT-2 was to be administered approximately 1 week later. The total number of PDT sessions per patient depended on response as follows: Complete responders (all lesions totally cleared clinically) 12 weeks after PDT-2: entered the FU part with no further treatment. Partial or non-responders 12 weeks after PDT-2 were retreated with by applying 2 additional PDTs in a second PDT cycle and then entered FU.
- Methyl-aminolevulinate: Topical application of methyl-aminolevulinate (MAL;160 mg/g). The dose of MAL was up to 1 g per PDT session (depending on size and number of target lesions located on neck, trunk, extremities, face or scalp, no more than 2 illumination areas with a maximum area incl. margin of 10cm², and a film thickness of about 1mm). Up to 4 administrations of study treatment (i.e. PDT sessions: drug application and subsequent illumination with BF-RhodoLED after 3h of drug incubation) were applied. For all patients, PDT-1 was to be administered directly after randomization and PDT-2 was to be administered approximately 1 week later. The total number of PDT sessions per patient depended on response as follows: Complete responders (all lesions totally cleared clinically) 12 weeks after PDT-2: entered the FU part with no further treatment. Partial or non-responders 12 weeks after PDT-2 were retreated by applying 2 additional PDTs in a second PDT cycle and then entered FU.
Period: Overall Study
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Started | 138 | 143
Completed (5 patients did not complete due to AE. In 3 of them these AEs were unrelated to study treatment.) | 128 | 132
Not Completed | 10 | 11
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Death | 0 | 1
Not completed — no visits 7 & 8/no visits after visit 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- BF-200 ALA: Topical application of BF-200 ALA gel (78 mg/g 5-aminolevulinic acid). The dose of BF-200 ALA was up to 1 g per PDT session (depending on size and number of target lesions located on neck, trunk, extremities, face or scalp, no more than 2 illumination areas with a maximum area incl. margin of 10cm², and a film thickness of about 1mm). Up to 4 administrations of study treatment (i.e. PDT sessions: drug application and subsequent illumination with BF-RhodoLED after 3h of drug incubation) were applied. For all patients, PDT-1 was to be administered directly after randomization and PDT-2 was to be administered approximately 1 week later. The total number of PDT sessions per patient depended on response as follows: Complete responders (lesions totally cleared clinically) 12 weeks after PDT-2: entered the FU part with no further treatment. Partial or non-responders 12 weeks after PDT-2 were retreated with by applying 2 additional PDTs in a second PDT cycle and then entered FU.
- Methyl-aminolevulinate: Topical application of methyl-aminolevulinate (MAL;160 mg/g). The dose of MAL was up to 1 g per PDT session (depending on size and number of target lesions located on neck, trunk, extremities, face or scalp, no more than 2 illumination areas with a maximum area incl. margin of 10cm², and a film thickness of about 1mm). Up to 4 administrations of study treatment (i.e. PDT sessions: drug application and subsequent illumination with BF-RhodoLED after 3h of drug incubation) were applied. For all patients, PDT-1 was to be administered directly after randomization and PDT-2 was to be administered approximately 1 week later. The total number of PDT sessions per patient depended on response as follows: Complete responders (lesions totally cleared clinically) 12 weeks after PDT-2: entered the FU part with no further treatment. Partial or non-responders 12 weeks after PDT-2 were retreated by applying 2 additional PDTs in a second PDT cycle and then entered FU.
- Total: Total of all reporting groups
Arm/Group | BF-200 ALA | Methyl-aminolevulinate | Total
Number analyzed (Participants) | 138 | 143 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 54 | 106
  >=65 years | 86 | 89 | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 68 | 122
  Male | 84 | 75 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 138 | 142 | 280
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Complete Response Rate Assessed 12 Weeks After the Last PDT
Description: Overall patient complete response rate assessed 12 weeks after the last PDT. The indicated values give the percentage of overall complete responders. An overall complete responder is defined as a patient in whom all treated lesions were cleared. The PP set is the primary analysis set for the analyses of the primary endpoint.
Time Frame: 12 weeks after the last PDT (please note: 2 PDT cycles, each cycle consisting of 2 PDTs (= maximum of 4 PDTs per patient) was possible).
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 121 | 110
Percentage of Patients | 93.4 [87.0 to 96.9] | 91.8 [84.6 to 96.0]
Statistical Analysis 1: Comparison: BF-200 ALA vs Methyl-aminolevulinate; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of -15%; p < 0.0001, Farrington and Manning Test; Difference of proportions; Difference in Percentage = 1.6, 97.5% CI 1-sided [lower limit -6.5]

2. Secondary Outcome: Lesion Complete Response Assessed 12 Weeks After the Last PDT
Description: Lesion complete response (completely cleared individual lesions) assessed 12 weeks after the last PDT. The indicated values give percentage of overall completely cleared individual lesions. The PP set is the primary analysis set for the analysis of the secondary endpoint.
Time Frame: as for outcome 1
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Individual Lesions
Units Other Than Participants: individual lesions
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 121 | 110
Number analyzed (individual lesions) | 148 | 127
Percentage of Individual Lesions | 94.6 [89.3 to 97.5] | 92.9 [86.6 to 96.5]

3. Secondary Outcome: Reduction of Lesion Area 12 Weeks After the Last PDT Compared to Baseline
Description: Reduction of total lesion area (summation of sizes of all treated lesions) per patient, assessed 12 weeks after the last PDT. The PP set is the primary analysis set for the analysis of the secondary endpoint.
  Please note that the high SD for BF-200 ALA is due to a patient who had increased lesion area fom 63 mm² at baseline to 225 mm² 12 weeks after PDT. This lesion area included a lesion that was later confirmed to be benign skin condition (lentigo solaris).
Time Frame: as for outcome 1
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 121 | 110
Percentage of Change | -94.5 (35.07) | -97.0 (13.37)

4. Secondary Outcome: Patient Complete Response 12 Weeks After PDT-2
Description: Patient complete response (complete clearance of all treated lesions) assessed 12 weeks after PDT-2 (first PDT cycle). The PP set is the primary analysis set for the analysis of the secondary endpoint.
Time Frame: 12 weeks after PDT-2 (=PDT cycle 1; please note: in this study 2 PDT cycles, each cycle consisting of 2 PDTs (= maximum of 4 PDTs per patient) was possible).
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 121 | 110
Percentage of Patients | 57.9 [48.5 to 66.7] | 56.4 [46.6 to 65.7]

5. Secondary Outcome: Cosmetic Outcome 12 Weeks After Last PDT (Including Patients With a Sum Score of 0 at Baseline)
Description: Overall cosmetic outcome 12 weeks after last PDT is calculated as difference between 12 weeks after PDT sum score and baseline sum score of all skin quality assessments. Each of the below skin quality characteristics are assessed on a 4-point scale from 0 (none) to 3 (severe) by the investigator at baseline and 12 weeks after last PDT:
  * Skin surface
  * Hyperpigmentation
  * Hypopigmentation
  * Mottled or irregular pigmentation
  * Degree of scarring
  * Atrophy
  Cosmetic outcome categories are:
  * Very good: 12 weeks sum score improved by at least 2 points compared to baseline
  * Good: 12 weeks sum score improved by 1 point compared to baseline
  * Satisfactory: 12 weeks sum score identical to the one at baseline
  * Unsatisfactory: 12 weeks sum score worsened by 1 point compared to baseline
  * Impaired: 12 weeks sum score worsened by at least 2 points compared to baseline
Time Frame: as for outcome 1
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 120 | 109
Percentage of Patients
  Very good | 23.3 [16.3 to 32.1] | 14.7 [8.9 to 23.0]
  Good | 11.7 [6.8 to 19.1] | 18.3 [11.8 to 27.2]
  Satisfactory | 35.8 [27.4 to 45.2] | 29.4 [21.2 to 39.0]
  Unsatisfactory | 14.2 [8.7 to 22.0] | 20.2 [13.3 to 29.2]
  Impaired | 15.0 [9.4 to 22.9] | 17.4 [11.1 to 26.1]

6. Secondary Outcome: Cosmetic Outcome 12 Weeks After the Last PDT (Including Patients With a Baseline Sum Score >1)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Per-protocol (PP) analysis set: All patients of the FAS without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 70 | 74
Percentage of Patients
  Very good | 40.0 [28.7 to 52.4] | 21.6 [13.2 to 33.0]
  Good | 20.0 [11.7 to 31.6] | 27.0 [17.7 to 38.8]
  Satisfactory | 22.9 [14.0 to 34.7] | 32.4 [22.3 to 44.4]
  Unsatisfactory | 11.4 [5.4 to 21.8] | 12.2 [6.1 to 22.3]
  Impaired | 5.7 [1.8 to 14.7] | 6.8 [2.5 to 15.7]

7. Other Pre Specified Outcome: Patient Recurrence Rate (Overall, Cumulative)
Description: Patient recurrence rate defined as the number of patients with at least one recurrent lesion during FU after complete clearance 12 weeks after the last PDT
Time Frame: 6, 12, 24, 36 and 60 months post-PDT
Population: Per protocol analysis set in the follow-up (PPS-FUP): all patients of the full analysis set in the follow-up (FAS-UP) without any major protocol deviations
Measure: Number; unit: percentage of patients (cumulative)
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 83 | 71
percentage of patients (cumulative) | 16.9 | 15.5

8. Other Pre Specified Outcome: Lesion Recurrence Rate (Cumulative)
Description: Lesion recurrence rate defined as the number of completely cleared lesions 12 weeks after the last PDT showing recurrence during FU. Overall and subgroup analysis (nodular basal cell carcinoma (nBCC) and superficial basal cell carcinoma (sBCC)).
Time Frame: 6, 12, 24, 36 and 60 months post-PDT
Population: Per protocol analysis in follow-up (PPS-FUP): All lesions in patients in the full analysis set in follow-up (FAS-FUP) without any major protocol deviations
Measure: Number; unit: percentage of lesions (cumulative)
Units Other Than Participants: Lesions
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
Number analyzed (Participants) | 83 | 71
Number analyzed (Lesions) | 104 | 82
percentage of lesions (cumulative)
  Overall | 13.5 | 13.4
  sBCC: number analyzed (Lesions) | 87 | 67
  sBCC | 10.3 | 11.9
  nBCC: number analyzed (Lesions) | 16 | 14
  nBCC | 25 | 21.4

ADVERSE EVENTS:
Time Frame: Each subject was assessed for a maximum of approximately 6 months after randomization depending on whether they received a second PDT cycle or not. Complete responders after the first PDT cycle were assessed for approximately 3 months after randomization. Additionally, there was a pre-randomization period of max. 2 weeks per patient.
Arm/Group | BF-200 ALA | Methyl-aminolevulinate
All-Cause Mortality (participants affected / at risk) | 0/138 | 1/143
Serious Adverse Events (participants affected / at risk) | 3/138 | 7/143
Other Adverse Events (participants affected / at risk) | 138/138 | 143/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=138) | Methyl-aminolevulinate (N=143)
Supraventricular trachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=138) | Methyl-aminolevulinate (N=143)
Application site pain (General disorders) | 134 (718) | 143 (751)
Application site erythema (General disorders) | 120 (309) | 126 (288)
Application site pruritus (General disorders) | 59 (91) | 49 (84)
Application site oedema (General disorders) | 42 (86) | 52 (108)
Application site paraesthesia (General disorders) | 40 (64) | 39 (65)
Application site scab (General disorders) | 34 (45) | 41 (49)
Application site induration (General disorders) | 32 (63) | 27 (50)
Application site discharge (General disorders) | 24 (38) | 24 (32)
Application site exfoliation (General disorders) | 22 (25) | 12 (13)
Application site erosion (General disorders) | 18 (22) | 9 (10)
Application site vesicles (General disorders) | 10 (13) | 11 (13)
Application site discolouration (General disorders) | 4 (4) | 8 (10)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (11)
Nasopharyngitis (Infections and infestations) | 11 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor will review results communications prior to public release and has to approve in order to ensure the adequate reporting of study results. The sponsor can't refuse publication for unfair reasons.